CLINICAL TRIAL: NCT06223217
Title: Development and Validation of the Modified Version of VascuQol Scale in Patients With Lower Extremity Peripheral Arterial Disease.
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); First Affiliated Hospital of Zhejiang University (Other); First People's Hospital of Hangzhou (Other); Huashan Hospital (Other); Hospital of Chengdu University of TCM (Unknown)
Responsible Party: Sponsor
Other Study IDs: VQL Study
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experiment group: Patients who undergoing endoluminal treatment for lower extremity peripheral arterial disease will complete the Modified version of the VascuQoL scale, the Chinese version of the VascuQoL scale, EQ-5D-5L Scale and the ABI test according to follow-up plan.
  Interventions: Other: Surveys and Questionnaires

INTERVENTIONS:
Other: Surveys and Questionnaires — The intervention consists of completing the Chinese version of Vascu-QoL scale and the modified version of Vascu-QoL scale

SUMMARY:
The purpose of this study is to assess the utility of the Modified version of VascuQol Scale as an effective biopsychosocial assessment tool for patients suffering from lower extremity peripheral arterial disease.

DETAILED DESCRIPTION:
In the prior study, the original 25-item VascuQol Scale demonstrates the limitation of dimensional mixing. As a result, we suggest improving the original scale by integrating the five dimensions and simplifying the objects. 480 patients will be recruited to complete the Chinese version of VascuQol Scale and the modified version. Reliability, validity, responsiveness, and diagnostic accuracy for CLTI will be used to evaluate whether the modified scale could serve as an effective biopsychosocial assessment tool for patients suffering from lower extremity peripheral arterial disease.

Study Procedures :

After signing the informed consent form, eligible patients and/or their legal guardians will complete the questionnaires.

Outcome measures:

Patient-Reported Outcomes via specific questionnaires

Participant numbers:

480 patients will be recruited

Data management:

Data will be collected directly from the patients. All paper patient records will be kept in locked filing cabinet. Electronic files will be saved on password protected folder

Oversight :

i) Data will be collected in a electric database; ii) all documents containing the identity of the participating subjects (non-objection, list of correspondence, etc.) will be kept away from personal data; iii) If it is a computerized document, it will be kept on the center's information server with access control by password.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-90
2. The patient is diagnosed with lower extremity peripheral arterial disease
3. The patient is willing to comply with specified follow-up evaluations at the specified times
4. The patient understands the nature of the procedure and provides written informed consent before enrolment in the study
5. Before enrolment, the guidewire has crossed the target lesion
6. No restrictions on Rutherford grading, TASC grading, GLASS grading

Exclusion Criteria:

1. Pregnant women or Female patients with potential childbearing
2. The patient is currently participating in another investigational drug or device study that has not reached the primary endpoint.
3. Patients unwilling or refusing to sign informed consent
4. Patients with other diseases that may seriously affect the quality of life, such as tumors, severe liver disease, cardiac insufficiency, etc., or those with a life expectancy of less than 2 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient is diagnosed with lower extremity peripheral arterial disease and no restrictions on Rutherford grading, TASC grading, GLASS grading.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the Modified version of VascuQol Scale | pre-operation；1-month；3-month；6-month；12-month
  It is one of the frequently used scales to measure quality of life in patients with lower extremity arterial disease. It evaluates 5 different categories such as the symptom, social, activity, pain and emotional with a total of 25 sub-items. A 7-point Likert system is used to score this scale. It is sufficient for each item to check the corresponding boxes. In Modified version，we adjusted the questionnaire items and structure based on the the Chinese version and results of the previous reserach.
the Chinese version of VascuQol Scale | pre-operation；1-month；3-month；6-month；12-month
  It is one of the frequently used scales to measure quality of life in patients with lower extremity arterial disease. It evaluates 5 different categories such as the symptom, social, activity, pain and emotional with a total of 25 sub-items. A 7-point Likert system is used to score this scale. It is sufficient for each item to check the corresponding boxes. In Chinese version，not only did we complete cultural adaptation, but we used the emoji-based visual analogue scale to help patients fill out the scales.

SECONDARY OUTCOMES:
Ankle brachial index（ABI） | pre-operation；6-month；12-month
  The ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium). Compared to the arm, lower blood pressure in the leg suggests blocked arteries due to peripheral artery disease (PAD). The ABPI is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure in the arm.
EQ-5D-5L Scale | pre-operation；1-month；3-month；6-month；12-month
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China